CLINICAL TRIAL: NCT05091307
Title: A Randomized, Double-blind, Phase 3 Study to Evaluate Safety, Reactogenicity, and Immunogenicity of Co-administration of Ad26.COV2.S and Influenza Vaccines in Healthy Adults 18 Years of Age and Older
Brief Title: A Study of Ad26.COV2.S and Influenza Vaccines in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109083; 2021-003953-43 (EudraCT Number); VAC31518COV3005 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-10-01; First posted 2021-10-25 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Prevention
MeSH Terms: interventions — Ad26COVS1; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-dose (SD) Influenza Vaccine and Placebo (Experimental): Participants aged greater than or equal to (>=) 18 years will receive a single intramuscular (IM) injection of Ad26.COV2.S and a seasonal Q SD influenza vaccine on Day 1 and placebo on Day 29.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo; Biological: Influenza Vaccine
- Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S (Placebo Comparator): Participants aged >=18 years will receive a single IM injection of placebo and a seasonal Q SD influenza vaccine on Day 1 followed by Ad26.COV2.S on Day 29.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo; Biological: Influenza Vaccine
- Group 3: Ad26.COV2.S + Q High-dose (HD) Influenza Vaccine and Placebo (Experimental): Participants aged >=65 years will receive a single IM injection of Ad26.COV2.S and a seasonal Q HD influenza vaccine on Day 1 followed by placebo on Day 29.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo; Biological: Influenza Vaccine
- Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S (Placebo Comparator): Participants aged >=65 years will receive a single IM injection of placebo and a seasonal Q HD influenza vaccine on Day 1 followed by Ad26.COV2.S on Day 29.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo; Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S will be administered as an IM injection.
  Other Names: VAC31518; JNJ-78436735
Other: Placebo — Placebo will be administered as an IM injection.
Biological: Influenza Vaccine — Influenza vaccine high and standard dose will be administered as IM injection.

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority (NI) of the humoral immune response of the 4 influenza vaccine strains after concomitant administration of the Ad26.COV2.S vaccine and a seasonal quadrivalent standard-dose influenza vaccine versus the administration of a seasonal quadrivalent standard-dose influenza vaccine administered alone; and to demonstrate the NI of the binding antibody response after concomitant administration of Ad26.COV2.S vaccine and a seasonal quadrivalent standard-dose influenza vaccine versus the administration of Ad26.COV2.S vaccine administered alone.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus(-2) (SARS CoV-2) is a highly transmissible and pathogenic coronavirus that has spread rapidly and globally and Influenza is a worldwide public health problem, responsible for significant morbidity and mortality. Ad26.COV2.S (also known as VAC31518, JNJ-78436735) is a monovalent vaccine composed of a recombinant, replication-incompetent human adenovirus type 26 (Ad26) vector, constructed to encode SARS-CoV-2 spike (S) protein, stabilized in its prefusion conformation. The seasonal influenza vaccines to be used in this study are quadrivalent (standard dose) and quadrivalent (high-dose) or equivalent formulated. The aim is to demonstrate the concomitant administration of the Ad26.COV2.S vaccine and a seasonal quadrivalent influenza vaccine (standard-dose) is non-inferior than the administration of either seasonal quadrivalent influenza vaccine (standard-dose) alone as measured by HI titers against each of the 4 influenza vaccine strains at 28 days after the administration of a quadrivalent seasonal influenza vaccine or Ad26.COV2.S vaccine alone as measured by Spiked-Enzyme-linked Immunosorbent Assay (S-ELISA) antibody titers at 28 days after the administration of the Ad26.COV2.S vaccine. This study consists of 3 phases: screening phase (Day -28 to 1), treatment phase (vaccination visits on Days 1 and 29), and a follow-up phase (28 days after each vaccination). Some of safety assessments will include physical examination, vital signs, clinical safety laboratory assessments, pregnancy testing, monitoring of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI). The total duration of the study is up to 7-8 months.

Note: The Informed Consent Form dated 25-Mar-2022 is final version of the study MASTER ICF, used by local countries to prepare the local language version of the ICF, which have been approved by the Ethics Committees. And the highlighted text in the ICF document are the guidance for country specific adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, and vital signs performed at screening. Participants may have underlying illnesses, as long as the symptoms and signs are medically controlled
* Participant either received complete primary vaccination with an authorized/licensed coronavirus disease-2019 (COVID-19) vaccine (completed greater than or equal to [>=] 6 months prior to the last vaccination received against COVID-19) or is COVID-19 vaccine-naive
* All participants who were born female and are of childbearing potential must: a. Have a negative highly sensitive urine pregnancy test at screening, b. Have a negative highly sensitive urine pregnancy test on the day of vaccination prior to each study vaccine administration
* Participant agrees to not donate or receive bone marrow, blood, and blood products from the administration of the study vaccine until 3 months after receiving the study vaccines
* Participant must be willing to provide verifiable identification to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancies considered cured with minimal risk of recurrence per investigator's clinical judgment)
* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature >= 38.0 degrees celsius (ºC) (100.4 degrees fahrenheit [°F]) within 24 hours prior to the planned dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator
* Participant has history of thrombosis with thrombocytopenia syndrome (TTS) or heparin-induced thrombocytopenia and thrombosis (HITT)
* Participant has history of capillary leak syndrome
* Participant received a licensed/registered severe acute respiratory syndrome coronavirus(-2) (SARS-CoV-2) vaccine less than 6 months prior to first study vaccination (other than study vaccination)
* Participant has a history of any neurological disorders or seizures including Guillain-Barre syndrome, with the exception of febrile seizures during childhood

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (31):
- United States (17):
  - Fiel Family and Sports Medicine Clinical Research Advantage, Tempe, Arizona
  - Wr McCr Llc, San Diego, California
  - Clinical Research of South Florida, an AMR Company, Coral Gables, Florida
  - AMR Fort Myers Clinical Physiology Associates, an AMR company, Fort Myers, Florida
  - Office of Emilio Mantero-Atienza, MD, Miami, Florida
  - University of Miami Health System, Miami, Florida
  - Premier Research Associate, Inc, Miami, Florida
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - I.D. Care, Inc., Hillsborough, New Jersey
  - Rochester Clinical Research, Inc, Rochester, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Ventavia Research Group, LLC, Keller, Texas
  - Research Your Health, Plano, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
- Belgium (4):
  - Anima, Alken
  - Institute of Tropical Medicine Antwerp, Antwerp
  - Clinical Pharmacology Unit, Merksem
  - Private Practice RESPISOM Namur, Namur
- Poland (10):
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Gdanskie Centrum Zdrowia, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdynia, Gdynia
  - Synexus Polska Sp z o o Oddzial w Katowicach, Katowice
  - Synexus Polska Sp Z O O Oddzial W Lodzi, Lodz
  - Synexus Polska Sp. z.o.o. Oddzial w Poznaniu, Poznan
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Synexus Polska Sp z o o Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp z o o Oddzial we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Tapia-Calle G, Aguilar G, Vaissiere N, Truyers C, Ylisastigui P, Buntinx E, Le Gars M, Struyf F, Scheper G, Douoguih M, Ruiz-Guinazu J; COV3005 Study group. Safety, reactogenicity, and immunogenicity of Ad26.COV2.S co-administered with a quadrivalent standard-dose or high-dose seasonal influenza vaccine: a non-inferiority randomised controlled trial. EClinicalMedicine. 2025 Jan 7;79:103016. doi: 10.1016/j.eclinm.2024.103016. eCollection 2025 Jan. PMID 39866854

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo: Participants aged greater than or equal to (>=) 18 years and older received a single intramuscular (IM) injection of Ad26.COV2.S at 5*10^10 viral particles (vp) dose level and a seasonal Q SD influenza vaccine with 60 micrograms (mcg) hemagglutinin (HA) on Day 1 followed by a single IM injection of placebo (matched to Ad26.COV2.S) on Day 29.
- Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S: Participants aged >=18 years and older received a single IM injection of placebo (matched to Ad26.COV2.S) and a seasonal Q SD influenza vaccine with 60 mcg of HA on Day 1 followed by a single IM injection of Ad26.COV2.S at 5*10^10 vp dose level on Day 29.
- Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo: Participants aged >=65 years and older received a single IM injection of Ad26.COV2.S at 5*10^10 vp dose level and a seasonal Q HD influenza vaccine with 240 mcg HA on Day 1 followed by a single IM injection of placebo (matched to Ad26.COV2.S) on Day 29.
- Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S: Participants aged >=65 years and older received a single IM injection of placebo (matched to Ad26.COV2.S) and a seasonal Q HD influenza vaccine with 240 mcg of HA on Day 1 followed by a single IM injection of Ad26.COV2.S at 5*10^10 vp dose level on Day 29.
Period: Overall Study
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Started (Randomized participants) | 382 | 386 | 47 | 46
Treated (Vaccinated participants) | 382 | 384 | 47 | 46
Completed | 312 | 316 | 43 | 44
Not Completed | 70 | 70 | 4 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 33 | 33 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 16 | 0 | 1
Not completed — Covid-19 Vaccine/Treatment | 14 | 15 | 1 | 1
Not completed — Initiated Prohibited Medication | 1 | 0 | 0 | 0
Not completed — Other | 4 | 4 | 0 | 0
Not completed — Randomized but not vaccinated | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants with a vaccine administration documented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S | Total
Number analyzed (Participants) | 382 | 384 | 47 | 46 | 859
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 336 | 337 | 0 | 0 | 673
  >=65 years | 46 | 47 | 47 | 46 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.92) | 45.5 (15.25) | 71.1 (4.58) | 71.3 (5.29) | 48.6 (16.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 177 | 22 | 33 | 423
  Male | 191 | 207 | 25 | 13 | 436
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 109 | 4 | 4 | 234
  Not Hispanic or Latino | 262 | 274 | 43 | 42 | 621
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 0 | 4
  Asian | 7 | 10 | 1 | 1 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 48 | 52 | 0 | 0 | 100
  White | 311 | 310 | 46 | 45 | 712
  More than one race | 9 | 3 | 0 | 0 | 12
  Unknown or Not Reported | 6 | 5 | 0 | 0 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 24 | 26 | 25 | 24 | 99
  Poland | 52 | 51 | 8 | 3 | 114
  United States | 306 | 307 | 14 | 19 | 646

OUTCOME MEASURES:

1. Primary Outcome: Groups 1 and 2: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibodies Against Each of the Four Influenza Vaccine Strains 28 Days After the Administration of a Seasonal Quadrivalent Standard-dose Influenza Vaccine
Description: GMTs of HI antibodies were measured using hemagglutination inhibition (HAI) assay against each of four influenza vaccine strains (A/Victoria [H1N1], A/Cambodia [H3N2], B/Victoria [B/Victoria] and B/Phuket [B/Yamagata]). This outcome measure was planned to be analyzed for specified arms only. PPII=Per-protocol influenza immunogenicity.
Time Frame: 28 days after vaccination with seasonal quadrivalent standard-dose influenza vaccine (Day 29)
Population: The PPII set included all randomized participants who received Ad26.COV2.S vaccine in combination with seasonal influenza vaccine for co-administration group and those who received seasonal influenza vaccine alone for control group, for whom immunogenicity data were available for at least one of influenza strains in vaccine. Participants with major protocol deviation were excluded from PPII analysis. 'N' (number of participants analyzed)=participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 320 | 333
Titers
  A/Victoria (H1N1) | 306 [271 to 346] | 393 [348 to 445]
  A/Cambodia (H3N2) | 134 [119 to 150] | 165 [147 to 186]
  B/Victoria (B/Victoria) | 38 [34 to 43] | 38 [33 to 43]
  B/Phuket (B/Yamagata) | 32 [29 to 36] | 33 [30 to 37]
Statistical Analysis 1: Comparison: Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo vs Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S; A/Victoria (H1N1): Based on analysis of variance (ANOVA) models, CIs around the difference (Group 2 [control group] minus Group 1 [CoAd group]) was calculated and back-transformed (by exponentiation: 2^CI) to CIs around a geometric mean ratio (GMR: GMTControl/GMTCoAd); Test type: Non-Inferiority — The criterion for non-inferiority (NI) was the upper bound of the 2-sided 95% CI for the GMR was below 1.5; ANOVA; Geometric Mean Ratio = 1.28, 95% CI 2-sided [1.09 to 1.53]
Statistical Analysis 2: Comparison: Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo vs Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S; A/Cambodia (H3N2): Based on analysis of variance (ANOVA) models, CIs around the difference (Group 2 [control group] minus Group 1 [CoAd group]) was calculated and back-transformed (by exponentiation: 2^CI) to CIs around a geometric mean ratio (GMR: GMTControl/GMTCoAd); Test type: Non-Inferiority — The criterion for NI was the upper bound of the 2-sided 95% CI for the GMR was below 1.5; ANOVA; Geometric Mean Ratio = 1.23, 95% CI 2-sided [1.05 to 1.45]
Statistical Analysis 3: Comparison: Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo vs Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S; B/Victoria (B/Victoria): Based on analysis of variance (ANOVA) models, CIs around the difference (Group 2 [control group] minus Group 1 [CoAd group]) was calculated and back-transformed (by exponentiation: 2^CI) to CIs around a geometric mean ratio (GMR: GMTControl/GMTCoAd); Test type: Non-Inferiority — The criterion for NI was the upper bound of the 2-sided 95% CI for the GMR was below 1.5; ANOVA; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.84 to 1.19]
Statistical Analysis 4: Comparison: Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo vs Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S; B/Phuket (B/Yamagata): Based on analysis of variance (ANOVA) models, CIs around the difference (Group 2 [control group] minus Group 1 [CoAd group]) was calculated and back-transformed (by exponentiation: 2^CI) to CIs around a geometric mean ratio (GMR: GMTControl/GMTCoAd); Test type: Non-Inferiority — The criterion for NI was the upper bound of the 2-sided 95% CI for the GMR was below 1.5; ANOVA; Geometric Mean Ratio = 1.03, 95% CI 2-sided [0.88 to 1.21]

2. Primary Outcome: Groups 1 and 2: Geometric Mean Concentrations (GMCs) of Antibodies Measured by Spiked-Enzyme-linked Immunosorbent Assay (S-ELISA) 28 Days After Administration of Ad26.COV2.S Vaccine
Description: GMCs of antibody titers measured by S-ELISA at 28 days after administration of Ad26.COV2.S vaccine was reported. This outcome measure was planned to be analyzed for specified arms only. Seronegative participants (at Day 1) who became serology positive during the study, participants with positive molecular test for severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) and major protocol deviation were excluded from PPSI analysis.
Time Frame: 28 days after vaccination with Ad26.COV2.S vaccine (Group 1: Day 29, Group 2: Day 57)
Population: The per protocol SARS-CoV-2 immunogenicity set (PPSI) included all randomized participants who received Ad26.COV2.S vaccine in combination with seasonal influenza vaccine for co-administration group and Ad26.COV2.S vaccine alone for control group, and for whom immunogenicity data was available. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Unit per milliliter (EU/mL)
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 257 | 209
ELISA Unit per milliliter (EU/mL) | 22531 [20140 to 25205] | 25035 [22189 to 28246]
Statistical Analysis 1: Comparison: Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo vs Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S; Based on analysis of variance (ANOVA) models, CIs around the difference (Group 2 [control group] minus Group 1 [CoAd group]) was calculated and back-transformed (by exponentiation: 2^CI) to CIs around a geometric mean ratio (GMR: GMTControl/GMTCoAd); Test type: Non-Inferiority — The criterion for NI was the upper bound of the 2-sided 95% CI for the GMR was below 1.5; ANOVA; Geometric Mean Ratio = 1.11, 95% CI 2-sided [0.97 to 1.26]

3. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) up to 7 Days After Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included erythema, swelling/induration, and pain/tenderness.
Time Frame: 7 days after first vaccination on Day 1 (up to Day 8); 7 days after second vaccination on Day 29 (up to Day 36)
Population: The full analysis set (FAS) included all randomized participants with at least 1 documented study vaccine administration. Here, 'n' (number analyzed) signifies participants who were evaluated at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants
  After first vaccination | 261 | 204 | 23 | 21
  After second vaccination: number analyzed (Participants) | 342 | 348 | 46 | 45
  After second vaccination | 34 | 210 | 3 | 24

4. Secondary Outcome: Number of Participants With Solicited Systemic AEs up to 7 Days After Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs included fever (defined as body temperature of 38.0-degree celsius or higher), headache, fatigue, myalgia, nausea, vomiting were collected within 7 days after each vaccination.
Time Frame: 7 days after first vaccination on Day 1 (up to Day 8); 7 days after second vaccination on Day 29 (up to Day 36)
Population: The FAS included all randomized participants with at least 1 documented study vaccine administration. Here, 'n' (number analyzed) signifies participants who were evaluated at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants
  After first vaccination | 256 | 205 | 30 | 26
  After second vaccination: number analyzed (Participants) | 342 | 348 | 46 | 45
  After second vaccination | 84 | 208 | 8 | 22

5. Secondary Outcome: Number of Participants With Unsolicited AEs up to 28 Days After Each Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after first vaccination on Day 1 (up to Day 29); 28 days after second vaccination on Day 29 (up to Day 57)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants
  After first vaccination | 71 | 71 | 10 | 9
  After second vaccination: number analyzed (Participants) | 342 | 348 | 46 | 45
  After second vaccination | 36 | 50 | 11 | 8

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. SAE was any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 12.5 months)
Population: The FAS included all randomized participants with at least 1 documented study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants | 9 | 7 | 1 | 2

7. Secondary Outcome: Number of Participants With Medically-attended Adverse Events (MAAEs)
Description: Number of participants with MAAEs was reported. MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. New onset of chronic diseases was collected as part of the MAAEs.
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 12.5 months)
Population: The FAS included all randomized participants with at least 1 documented study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants | 51 | 51 | 11 | 16

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with AESIs was reported. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, was considered to be an AESI in this study. A suspected TTS case was defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/microliter.
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 12.5 months)
Population: The FAS included all randomized participants with at least 1 documented study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants | 9 | 12 | 0 | 0

9. Secondary Outcome: Number of Participants With AEs Leading to Withdrawal From the Study
Description: Number of participants with AE leading to withdrawal from the study was reported.
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 12.5 months)
Population: The FAS included all randomized participants with at least 1 documented study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 382 | 384 | 47 | 46
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Groups 3 and 4: GMTs of HI Antibodies Against Each of the Four Influenza Vaccine Strains 28 Days After the Administration of a Seasonal Quadrivalent High-dose Influenza Vaccine
Description: GMTs of HI antibodies were measured using hemagglutination inhibition (HAI) assay against each of four influenza vaccine strains (A/Victoria [H1N1], A/Tasmania[H3N2], B/Washington [B/Victoria] and B/Phuket [B/Yamagata]). This outcome measure was planned to be analyzed for specified arms only.
Time Frame: 28 days after vaccination with seasonal quadrivalent high-dose influenza vaccine (Day 29)
Population: The PPII set included all randomized participants who received Ad26.COV2.S vaccine in combination with a seasonal influenza vaccine for the coadministration group and those who received a seasonal influenza vaccine alone for the control group, for whom immunogenicity data were available for at least one of the influenza strains in the vaccine. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 43 | 41
Titers
  A/Victoria (H1N1) | 286 [204 to 400] | 484 [369 to 636]
  A/Tasmania (H3N2) | 284 [200 to 402] | 509 [365 to 711]
  B/Washington (B/Victoria) | 61 [46 to 81] | 75 [53 to 106]
  B/Phuket (B/Yamagata) | 38 [29 to 50] | 39 [30 to 52]

11. Secondary Outcome: Group 3 and 4: GMCs of Antibodies Measured by S-ELISA 28 Days After Administration of Ad26.COV2.S Vaccine
Description: GMCs of antibody titers measured by S-ELISA at 28 days after administration of Ad26.COV2.S vaccine was reported. This outcome measure was planned to be analyzed for specified arms only. Seronegative participants (at Day 1) who became serology positive during the study, participants with positive molecular test for SARSCoV-2 and major protocol deviation were excluded from PPSI analysis.
Time Frame: 28 days after vaccination with Ad26.COV2.S vaccine (Group 3: Day 29, Group 4: Day 57)
Population: The PPSI included all randomized participants who received Ad26.COV2.S vaccine in combination with seasonal influenza vaccine for the co-administration group and Ad26.COV2.S vaccine alone for the control group, and for whom immunogenicity data was available. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 39 | 33
EU/mL | 17569 [13391 to 23051] | 20743 [12732 to 33794]

12. Secondary Outcome: GMCs of Antibodies Measured by S-ELISA 28 Days After Administration of Ad26.COV2.S Vaccine in COVID-19 Vaccine Naive Participants
Description: GMCs of antibodies measured by S-ELISA 28 days after administration of Ad26.COV.S vaccine in Covid-19 vaccine naive participants was reported. In the below data table, '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Time Frame: 28 days after the administration of Ad26.COV2.S vaccine (that is, for Groups 1 and 3: Day 29; for Groups 2 and 4: Day 57)
Population: PPSI included all randomized participants who received Ad26.COV2.S vaccine in combination with seasonal influenza vaccine for co-administration group and Ad26.COV2.S vaccine alone for control group and for whom immunogenicity data was available. Participants with positive molecular test for SARSCoV-2 were also excluded. Here, 'N'(number of participants analyzed)=who were evaluable for this outcome measure, 'n'(number analyzed)=participant who were evaluated at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 46 | 40 | 0 | 1
EU/mL | 10340 [6557 to 16306] | 14704 [9010 to 23998] |  | 38905 [NA to NA] — Here, 'NA' indicated that lower limit and upper limit of 95% confidence interval could not be estimated as only 1 participant was analyzed on Day 57 in Group 4.

13. Secondary Outcome: Percentage of Participants With Seroconversion for Each of the 4 Influenza Vaccine Strains at 28 Days After the Administration of a Seasonal Quadrivalent (High-dose and Standard-dose) Influenza Vaccine
Description: Seroconversion was defined for each of the 4 influenza vaccine strains (For group 1 and 2: A/Victoria [H1N1], A/Cambodia [H3N2], B/Victoria [B/Victoria], B/Phuket [B/Yamagata]; For group 3 and 4: A/Victoria [H1N1], B/Phuket (B/Yamagata), A/Tasmania [H3N2], B/Washington [B/Victoria]) at 28 days after the administration of a seasonal quadrivalent (high-dose and standard-dose) influenza vaccine: HI titer greater than or equal to (>=) 1:40 in participants with a pre-vaccination HI titer of less than (<) 1:10, or a >=4-fold HI titer increase in participants with a pre-vaccination HI titer of >= 1:10. In the below data table, '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Time Frame: 28 days after the administration of a seasonal quadrivalent influenza vaccine (Day 29)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 320 | 333 | 43 | 41
Percentage of participants
  A/Victoria (H1N1) | 64.1 [58.5 to 69.3] | 70.0 [64.7 to 74.8] | 65.1 [49.1 to 79.0] | 70.7 [54.5 to 83.9]
  A/Cambodia (H3N2): number analyzed (Participants) | 320 | 333 | 0 | 0
  A/Cambodia (H3N2) | 39.1 [33.7 to 44.6] | 46.8 [41.4 to 52.4] |  |
  B/Victoria (B/Victoria): number analyzed (Participants) | 320 | 333 | 0 | 0
  B/Victoria (B/Victoria) | 42.8 [37.3 to 48.4] | 43.5 [38.1 to 49.1] |  |
  B/Phuket (B/Yamagata) | 35.3 [30.1 to 40.8] | 36.9 [31.7 to 42.4] | 37.2 [23.0 to 53.3] | 34.1 [20.1 to 50.6]
  A/Tasmania (H3N2): number analyzed (Participants) | 0 | 0 | 43 | 41
  A/Tasmania (H3N2) |  |  | 72.1 [56.3 to 84.7] | 70.7 [54.5 to 83.9]
  B/Washington (B/Victoria): number analyzed (Participants) | 0 | 0 | 43 | 41
  B/Washington (B/Victoria) |  |  | 41.9 [27.0 to 57.9] | 53.7 [37.4 to 69.3]

14. Secondary Outcome: Percentage of Participants With Seroprotection for Each of the 4 Influenza Vaccine Strains as HI Titer >= 1:40 at 28 Days After the Administration of a Seasonal Quadrivalent (High-dose and Standard-dose) Influenza Vaccine
Description: Seroprotection was defined for each of the 4 influenza vaccine strains (For group 1 and 2: A/Victoria [H1N1], A/Cambodia [H3N2], B/Victoria [B/Victoria], B/Phuket [B/Yamagata]; For group 3 and 4: A/Victoria [H1N1], B/Phuket (B/Yamagata), A/Tasmania [H3N2], B/Washington [B/Victoria]) as HI titer >=1:40 at 28 days after the administration of a seasonal quadrivalent (high-dose and standard-dose) influenza vaccine. In the below data table, '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Time Frame: 28 days after the administration of a seasonal quadrivalent influenza vaccine (Day 29)
Population: The PPII set included all randomized participants who received Ad26.COV2.S vaccine in combination with seasonal influenza vaccine for coadministration group and those who received seasonal influenza vaccine alone for control group, for whom immunogenicity data were available for at least one of influenza strains in vaccine. Participants with major protocol deviation were excluded from PPII analysis. 'N' (number of participants analyzed)=participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
Number analyzed (Participants) | 320 | 333 | 43 | 41
Percentage of participants
  A/Victoria (H1N1) | 97.8 [95.5 to 99.1] | 97.3 [94.9 to 98.8] | 100.0 [91.8 to 100.0] | 100.0 [91.4 to 100.0]
  A/Cambodia (H3N2): number analyzed (Participants) | 320 | 333 | 0 | 0
  A/Cambodia (H3N2) | 92.8 [89.4 to 95.4] | 93.4 [90.2 to 95.8] |  |
  B/Victoria (B/Victoria): number analyzed (Participants) | 320 | 333 | 0 | 0
  B/Victoria (B/Victoria) | 56.9 [51.2 to 62.4] | 57.4 [51.8 to 62.7] |  |
  B/Phuket (B/Yamagata) | 52.2 [46.6 to 57.8] | 55.0 [49.4 to 60.4] | 62.8 [46.7 to 77.0] | 63.4 [46.9 to 77.9]
  A/Tasmania (H3N2): number analyzed (Participants) | 0 | 0 | 43 | 41
  A/Tasmania (H3N2) |  |  | 97.7 [87.7 to 99.9] | 100.0 [91.4 to 100.0]
  B/Washington (B/Victoria): number analyzed (Participants) | 0 | 0 | 43 | 41
  B/Washington (B/Victoria) |  |  | 79.1 [64.0 to 90.0] | 82.9 [67.9 to 92.8]

ADVERSE EVENTS:
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 12.5 months)
Description: The full analysis set (FAS) included all randomized participants with at least 1 documented study vaccine administration.
Arm/Group | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S
All-Cause Mortality (participants affected / at risk) | 0/382 | 0/384 | 1/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 9/382 | 7/384 | 1/47 | 2/46
Other Adverse Events (participants affected / at risk) | 45/382 | 45/384 | 11/47 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo (N=382) | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S (N=384) | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo (N=47) | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S (N=46)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Chronic Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0
Biliary Obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Optic Neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26.COV2.S + Quadrivalent (Q) Standard-Dose (SD) Influenza Vaccine and Placebo (N=382) | Group 2: Placebo + Q SD Influenza Vaccine and Ad26.COV2.S (N=384) | Group 3: Ad26.COV2.S + Q High Dose (HD) Influenza Vaccine and Placebo (N=47) | Group 4: Placebo + Q HD Influenza Vaccine and Ad26.COV2.S (N=46)
Covid-19 (Infections and infestations) | 42 | 42 | 10 | 5
Nasopharyngitis (Infections and infestations) | 3 | 5 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (3):
  • Study Protocol (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05091307/Prot_001.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT05091307/SAP_002.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT05091307/ICF_005.pdf